CLINICAL TRIAL: NCT00309465
Title: A Study of the Relationship Between the Proportional Insulin Glargine Evening Dose and the Perioperative Serum Glucose Values in Patients With Diabetes Undergoing Surgery
Brief Title: Perioperative Insulin Glargine Dosing Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tamra Dukatz (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor-Investigator, Tamra Dukatz, Principal Investigator, Corewell Health East
Organization: Corewell Health East (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HIC 2005-080
Record Dates: First submitted 2006-03-30; First posted 2006-03-31 (Estimated); Results first posted 2012-12-03 (Estimated); Last update posted 2012-12-03 (Estimated); Status verified 2012-11

CONDITIONS: Diabetes; Surgery
Keywords: Diabetes; Insulin Glargine; Surgery
MeSH Terms: conditions — Diabetes Mellitus | interventions — Insulin Glargine; Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Patients in Group 1 will administer 80% of their usual insulin glargine dose.
  Interventions: Drug: Lantus
- 2 (Active Comparator): Group 2 patients will contact their own diabetes care physician and follow those recommendations for the dose.
  Interventions: Other: Insulin
- 3 (Experimental): Group 3 patients will take 50%, 80%, or 100% of their usual insulin glargine dose. Which of those three percentages will be determined by the midpoint of the patient's usual self-reported fasting blood sugar (FBS) range and whether the patients is also taking a rapid-acting insulin.
  Interventions: Drug: Lantus

INTERVENTIONS:
Drug: Lantus — Patients in Group 1 will administer 80% of their usual insulin glargine dose.
  Other Names: Lantus, Insulin
  Arms: 1
Other: Insulin — Group 2 patients will contact their own diabetes care physician and follow those recommendations for the dose
  Other Names: As directed by regular physician
  Arms: 2
Drug: Lantus — Group 3 patients will take 50%, 80%, or 100% of their usual insulin glargine dose. Which of those three percentages will be determined by the midpoint of the patient's usual self-reported fasting blood sugar (FBS) range and whether the patients is also taking a rapid-acting insulin.
  Arms: 3

SUMMARY:
The main objective of this study is to compare three strategies of evening insulin glargine dosing to preoperative glucose values in patients with diabetes undergoing surgery to determine which dosing strategies most often achieves the admission target study values of 100-179 mg/dl.

DETAILED DESCRIPTION:
There are no evidence-based guidelines for insulin glargine (Lantus) dosing in the perioperative setting. Insulin glargine provides peakless 24-hour coverage of basal insulin needs for people with both Type 1 and Type 2 diabetes. Insulin glargine may be used as the sole insulin or in combination with other rapid-acting insulin to achieve glycemic control.

Anesthesia literature recommends that blood sugar values on insulin-dependent patients be maintained between 120-180 mg/dl in most surgeries. Symptoms of low blood sugar are undetectable in anesthetized patients, and blood glucose is tested at least hourly. Since patients are still awake and alert toward hypoglycemic symptoms in the preoperative area, the admission target study values are 100-179 mg/dl. Glucose values greater than 200 mg/dl have been associated with increased rates of infection, and exacerbated complications if a major cardiovascular event happens.

Frequently insulin glargine is administered in the evening. Patients who are scheduled for surgery in the morning are asked not to eat or drink after midnight. Some endocrinology experts recommend that all or part of the patient's usual insulin glargine should be given to avoid high blood sugar; however, whenever insulin is given without food, the possibility of low blood sugar exists.

1. Patients in Group 1 will administer 80% of their usual insulin glargine dose.
2. Group 2 patients will contact their own diabetes care physician and follow those recommendations for the dose.
3. Group 3 patients will take 50%, 80%, or 100% of their usual insulin glargine dose. Which of those three percentages will be determined by the midpoint of the patient's usual self-reported fasting blood sugar (FBS) range and whether the patients is also taking a rapid-acting insulin.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for Surgical Procedure
* Self Management of Diabetes
* Currently on Evening Insulin Glargine prescribed by Primary Care Physician
* Age 18 or over
* Able to Communicate Clearly over the Phone
* Pre-screened by Anesthesia Department > 48 hours prior to Surgery

Exclusion Criteria:

* On Glucocorticoid Medication
* On Insulin Glargine Dual Dosing or Sliding Scale Regimen
* History of Hypoglycemia Unawareness
* Pregnancy or Lactating Female
* On Insulin Glargine for < 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 402 (Actual)
Dates: Start 2005-10; Primary Completion 2008-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tamra Dukatz, MSN, CRNA, Principal Investigator — Corewell Health East
Locations (2):
- United States (2):
  - William Beaumont Hospital, Royal Oak, Michigan
  - William Beaumont Hospital, Troy, Michigan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment at William Beaumont Heath System Royal Oak and Troy campuses commenced in October 2005 and was completed in September 2008.
Pre-assignment Details: Subjects were stratified into groups (insulin glargine only group and insulin glargine plus bolus group) by the absence or presence of daily rapid-acting (or short-acting) insulin in regimen. The two groups were then randomized into Take 80%, Call Physician or Dose Table strategies. One subject was excluded from analysis due to eligibility error.
Groups:
- Take 80% (Insulin Glargine Only Group): Subjects were instructed to self-administer 80% of the usual insulin glargine dose on the evening before surgery.
- Call Physician (Insulin Glargine Only Group); Call Physician (Insulin Glargine Plus Bolus Group: Subjects were instructed to call their own physician for the insulin glargine dose to administer the evening before surgery.
- Dose Table (Insulin Glargine Only Group): Subjects were instructed to self-administer: (a) 50% of their usual insulin glargine if the midpoint of their usual self-reported fasting blood glucose value was < 150 mg/dl or (b) 80% of their usual insulin glargine if the midpoint of their usual self-reported fasting blood glucose range was > or = 150 mg/dl.
- Take 80% (Insulin Glargine Plus Bolus Group): Subjects were instructed to self-administer 80% of the usual insulin glargine dose the evening before surgery
- Dose Table (Insulin Glargine Plus Bolus Group): Subjects were instructed to self-administer: (a) 80% of the usual insulin glargine dose if the midpoint of self-reported usual fasting blood glucose value was <150 mg/dl or (b) 100% of the usual insulin glargine dose if the midpoint of the self-reported usual fasting blood glucose range was > or = 150 mg/dl.
Period: Overall Study
Arm/Group | Take 80% (Insulin Glargine Only Group) | Call Physician (Insulin Glargine Only Group) | Dose Table (Insulin Glargine Only Group) | Take 80% (Insulin Glargine Plus Bolus Group) | Call Physician (Insulin Glargine Plus Bolus Group | Dose Table (Insulin Glargine Plus Bolus Group)
Started | 58 | 58 | 58 | 76 | 76 | 76
Completed | 58 | 58 | 58 | 75 (One subject was excluded due to eligibility error.) | 76 | 76
Not Completed | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Call Physician (Insulin Glargine Only Group): Subjects were instructed to call their physician for the insulin glargine dose to administer the evening before surgery.
- Dose Table (Insulin Glargine Only Group): Subjects were instructed to self-administer: (a) 50% of their usual insulin glargine if the midpoint of their usual self-reported fasting blood glucose range was < 150 mg/dl or (b) 80% of their usual insulin glargine if the midpoint of their usual fasting blood glucose range was > or = 150 mg/dl.
- Dose Table (Insulin Glargine Plus Bolus Group): Subjects were instructed to self administer: (a) 80% of the usual insulin glargine dose if the midpoint of self-reported usual fasting blood glucose range was <150 mg/dl or (b) 100% of the usual insulin glargine dose if the midpoint of the self-reported usual fasting blood glucose range was > or = 150 mg/dl.
- Total: Total of all reporting groups
Arm/Group | Take 80% (Insulin Glargine Only Group) | Call Physician (Insulin Glargine Only Group) | Dose Table (Insulin Glargine Only Group) | Take 80% (Insulin Glargine Plus Bolus Group) | Call Physician (Insulin Glargine Plus Bolus Group | Dose Table (Insulin Glargine Plus Bolus Group) | Total
Number analyzed (Participants) | 58 | 58 | 58 | 75 | 76 | 76 | 401
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 37 | 34 | 31 | 52 | 53 | 52 | 259
  >=65 years | 21 | 24 | 27 | 23 | 23 | 24 | 142
Age Continuous [Mean (Standard Deviation); unit: years] | 60.1 (10.0) | 61.5 (11.4) | 63.1 (11.6) | 55.8 (15.9) | 58.4 (12.0) | 57.3 (13.3) | 59.1 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 27 | 28 | 43 | 41 | 38 | 207
  Male | 28 | 31 | 30 | 32 | 35 | 38 | 194
Region of Enrollment [Number; unit: participants]
  United States | 58 | 58 | 58 | 75 | 76 | 76 | 401

OUTCOME MEASURES:

1. Primary Outcome: Primary: Preoperative Fasting Blood Sugar Upon Arrival at the Hospital Prior to Surgery
Description: Venous blood glucose values were obtained in the preoperative nursing unit. Blood glucose values were analyzed for achievement of target 100-179 mg/dl range and extended 80-249 mg/dl range. Analyses were by intention to treat.
Time Frame: Day 1
Population: Percentage of subjects that achieved preoperative blood glucose value of 100-179 mg/dl and 80-249 mg/dl. Analyses were by intention to treat.
Measure: Number; unit: Percentage of subjects
Groups:
- Take 80% (Insulin Glargine Only Group): Subjects self-administered 80% of usual insulin glargine dose on the evening before surgery
- Call Physician (Insulin Glargine Only Group): Subjects called their own physicians for insulin glargine dose on the evening before surgery
- Dose Table (Insulin Glargine Only Group): Subjects administered: (a) 50% of their usual insulin glargine dose if midpoint of usual self-reported fasting blood glucose range was <150 mg/dl or (b) 80% of usual insulin glargine dose if midpoint of usual self-reported fasting blood glucose range was > or = 150 mg/dl
- Take 80% (Insulin Glargine Plus Bolus Group): Subjects self-administered 80% of the usual insulin glargine dose on the evening before surgery
- Call Physician (Insulin Glargine Plus Bolus Group: Subjects called their own physicians for the insulin glargine dose to administer on the evening before surgery
- Dose Table (Insulin Glargine Plus Bolus Group): Subjects administered: (a) 80% of their usual insulin glargine dose if the midpoint of self-reported usual fasting blood glucose range was <150 mg/dl or (b) 100% of their usual insulin glargine dose if midpoint of self-reported usual fasting blood glucose ragne was > or = 150 mg/dl
Arm/Group | Take 80% (Insulin Glargine Only Group) | Call Physician (Insulin Glargine Only Group) | Dose Table (Insulin Glargine Only Group) | Take 80% (Insulin Glargine Plus Bolus Group) | Call Physician (Insulin Glargine Plus Bolus Group | Dose Table (Insulin Glargine Plus Bolus Group)
Number analyzed (Participants) | 58 | 58 | 58 | 75 | 76 | 76
Percentage of subjects
  Achievement of 100-179 mg/dl | 58.6 | 72.4 | 74.1 | 58.7 | 52.6 | 63.2
  Achievement of 80-249 mg/dl | 89.7 | 89.7 | 98.3 | 81.3 | 81.6 | 93.4
Statistical Analysis 1: Comparison: Take 80% (Insulin Glargine Only Group) vs Call Physician (Insulin Glargine Only Group) vs Dose Table (Insulin Glargine Only Group); Comparison for Target Blood Glucose Achievement of 100-179 mg/dl; Test type: Superiority or Other; p = 0.332, Chi-squared — P-value for three dosing strategies in insulin glargine only group in fasting blood glucose achievement of 100-179 mg/dl range
Statistical Analysis 2: Comparison: Take 80% (Insulin Glargine Plus Bolus Group) vs Call Physician (Insulin Glargine Plus Bolus Group vs Dose Table (Insulin Glargine Plus Bolus Group); Comparison for Target Achievement of blood glucose values of 100-179 mg/dl; Test type: Superiority or Other; p = 0.294, Chi-squared — P value is for three strategies in insulin glargine plus bolus group for fasting blood glucose achievement of 100-179 mg/dl
Statistical Analysis 3: Comparison: Take 80% (Insulin Glargine Only Group) vs Call Physician (Insulin Glargine Only Group) vs Dose Table (Insulin Glargine Only Group); Comparison of Achievement of blood glucose values of 80-249 mg/dl; Test type: Superiority or Other; p = 0.162, Chi-squared — P value is for three strategies in insulin glargine only group for achievement of 80-249 mg/dl
Statistical Analysis 4: Comparison: Take 80% (Insulin Glargine Plus Bolus Group) vs Call Physician (Insulin Glargine Plus Bolus Group vs Dose Table (Insulin Glargine Plus Bolus Group); Comparison of Achievement of blood glucose values of 80-249 mg/dl; Test type: Superiority or Other; p = 0.031, Chi-squared — P value is for three strategies in insulin glargine plus bolus group in achievement of fasting blood glucose value of 80-249 mg/dl

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for the preoperative period on the day of surgery. Severe hyperglycemia resulting in surgery cancellation and severe hypoglycemia resulting in loss of consciousness were defined as severe adverse events.
Groups:
- Call Physician (Insulin Glargine Only Group): Subjects called physician for the insulin glargine dose on the evening before surgery.
- Dose Table (Insulin Glargine Only Group): Subjects administered: (a) 50% of usual insulin glargine dose if midpoint of usual self-reported fasting blood glucose <150 mg/dl or (b) 80% of usual insulin glargine dose if midpoint of usual self-reported fasting blood glucose > or =150 mg/dl
- Take 80% (Insuling Glargine Plus Bolus Group): Subjects self-administered 80% of usual insulin glargine dose on the evening before surgery
- Call Physician (Insulin Glargine Plus Bolus Group): Subjects called physician for the insulin glargine dose to administer on the evening before surgery.
- Dose Table (Insulin Glargine Plus Bolus Group): Subjects administered: (a) 80% of usual insulin glargine if midpoint of usual self-reported fasting blood glucose was <150 mg/dl or (b) 100% of usual insulin glargine dose if midpoint of usual self-reported fasting blood glucose was < or =150 mg/dl.
Arm/Group | Take 80% (Insulin Glargine Only Group) | Call Physician (Insulin Glargine Only Group) | Dose Table (Insulin Glargine Only Group) | Take 80% (Insuling Glargine Plus Bolus Group) | Call Physician (Insulin Glargine Plus Bolus Group) | Dose Table (Insulin Glargine Plus Bolus Group)
Serious Adverse Events (participants affected / at risk) | 0/58 | 1/58 | 0/58 | 0/75 | 0/76 | 0/76
Other Adverse Events (participants affected / at risk) | 1/58 | 0/58 | 0/58 | 1/75 | 0/76 | 1/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Take 80% (Insulin Glargine Only Group) (N=58) | Call Physician (Insulin Glargine Only Group) (N=58) | Dose Table (Insulin Glargine Only Group) (N=58) | Take 80% (Insuling Glargine Plus Bolus Group) (N=75) | Call Physician (Insulin Glargine Plus Bolus Group) (N=76) | Dose Table (Insulin Glargine Plus Bolus Group) (N=76)
Severe Hyperglycemia resulting in surgery cancellation (Metabolism and nutrition disorders) | 0 | 1 (1) | 0 | 0 | 0 | 0 — A subject with type 2 diabetes had inadvertently self-administered an overdose of rapid-acting insulin two days before surgery. Hypoglycemia treatment rendered and the basal insulin dose omitted that day leading to BG of 644 mg/dl on day of surgery.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Take 80% (Insulin Glargine Only Group) (N=58) | Call Physician (Insulin Glargine Only Group) (N=58) | Dose Table (Insulin Glargine Only Group) (N=58) | Take 80% (Insuling Glargine Plus Bolus Group) (N=75) | Call Physician (Insulin Glargine Plus Bolus Group) (N=76) | Dose Table (Insulin Glargine Plus Bolus Group) (N=76)
Moderate Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 1 — Blood glucose value between 40-59 mg/dl in preoperative area, without loss of consciousness
Severe hyperglycemia without surgery cancellation (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 — Blood glucose >400 mg/dl in preoperative area

LIMITATIONS AND CAVEATS:
Limitations include use of point-of-care glucometers, which are less precise than central laboratory testing; estimated 75% power in the insulin glargine only group; and varying fasting lengths, usual glycemic control and surgery starting times.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No